CLINICAL TRIAL: NCT03467906
Title: Role of Dietary Habits in Efficacy of Bariatric Surgery - Study B
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Frank AJL Scheer, PhD, Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2017P002526B; R01HL140574 (NIH)
Record Dates: First submitted 2018-03-12; First posted 2018-03-16 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Bariatric Surgery; Sleeve Gastrectomy; Obesity
Keywords: Diet; Dietary Habits; Weight changes
MeSH Terms: conditions — Obesity; Feeding Behavior; Body Weight Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, urine, saliva.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Weight loss < median of group: Sleeve gastrectomy surgery patients will take part in in-laboratory assessment. Based on 1-year post-surgical weight loss, a median split will be done to allocate subjects to one of two groups.
  Interventions: Other: In-laboratory assessment
- Weight loss > median of group: Sleeve gastrectomy surgery patients will take part in in-laboratory assessment. Based on 1-year post-surgical weight loss, a median split will be done to allocate subjects to one of two groups.
  Interventions: Other: In-laboratory assessment

INTERVENTIONS:
Other: In-laboratory assessment — Participants will stay in the laboratory for two days and one night during which they will complete questionnaires, have blood drawn, and have other measurements taken.

SUMMARY:
The purpose of the study is to compare dietary habits after bariatric surgery in patients with poor weight loss versus good weight loss outcomes.

DETAILED DESCRIPTION:
The obesity epidemic is a major public health concern with a significant economic burden in the USA. Bariatric surgery is the most effective and durable weight loss treatment, with long-term cardiometabolic health benefits. Among different types of bariatric procedures, sleeve gastrectomy (SG) has become the most commonly performed in USA. While SG is expected to result in a 50-60% excess weight loss, inter-individual differences in weight loss are large and approximately 25% of patients can be considered poor weight-loss responders who either do not lose a substantial amount of weight or regain the lost weight afterwards. The mechanisms underlying this clinical variation remain unknown and interventions to improve on these outcomes critically lacking. Of interest, altered daily dietary habits are experienced by a substantial proportion of bariatric surgery candidates, raising the question whether such alterations may contribute to inter-individual differences in weight loss success. Therefore, the purpose of the study is to compare dietary habits after bariatric surgery in patients with different weight loss outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Bariatric surgery (sleeve gastrectomy) patients

Exclusion Criteria:

* Insulin-dependent diabetes
* Anemia
* Smoking
* Shift work within the past 1 year
* Drug or alcohol dependency
* Bipolar disorder
* Post traumatic stress disorder (PTSD)

Ages: 22 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients that have undergone sleeve gastrectomy surgery.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Self-rated hunger | One day of laboratory protocol
  Hunger measured from the visual analogue scale (VAS) questionnaire

SECONDARY OUTCOMES:
Self-rated appetite | One day of laboratory protocol
  Appetite measured from the visual analogue scale (VAS) questionnaire
Appetite-regulating hormones | One day of laboratory protocol
  Appetite-regulating hormones from blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Frank Scheer, PhD, Principal Investigator — Brigham and Women's Hospital; Ali Tavakkoli, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No